CLINICAL TRIAL: NCT03391089
Title: Non-contact Intraoperative Optical Imaging During Spinal Procedures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Victor Yang, Senior Scientist, Physical Sciences Platform, Sunnybrook Health Sciences Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 406-2015
Record Dates: First submitted 2017-12-18; First posted 2018-01-05 (Actual); Last update posted 2018-01-05 (Actual); Status verified 2017-12

CONDITIONS: Computer-assisted Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BBL Experimental Navigation System (Experimental): As this is a single arm trial, all participants receive treatment.
  Interventions: Device: BBL Experimental Navigation System

INTERVENTIONS:
Device: BBL Experimental Navigation System — Comparison of accuracy of screw placement using experimental system.

SUMMARY:
Current spine procedures can suffer from a variety of complications resulting in a high incidence (up to 55%) of misplaced screws and implants. This can lead to devastating clinical consequences, including neurologic and vascular injury, and extensive physical, mental, and economic damage. Surgical navigation has a great potential to reduce these risks through accurate guidance; however present technologies rely on intraoperative imaging that uses ionizing radiation (e.g. computed tomography, or fluoroscopy), which limits surgical anatomy registration updates to less than 3-4 time points during surgery. They also require cumbersome and lengthy set-up and registration of fiducial markers and have limited abilities to account for motion that occurs during surgery and patient positioning. Therefore, the investigators propose a real-time intraoperative optical topographical imaging based surgical guidance system capable of accurately guiding the placement of implanted devices such as screws.

DETAILED DESCRIPTION:
The hypothesis is that optical visualization of surgically exposed anatomy with the Biophotonics and Bioengineering Laboratory (BBL) surgical navigation prototype, when registered with pre-operative imaging (CT or MRI), can accurately estimate subsurface anatomy and allow tracking the position of surgical instruments in real-time, using an intraoperative non-contact optical imaging system during spinal surgical procedures. This is based on the completed preliminary study of 40 spinal procedures. The specific research aim is as follows: Validate the ability of the BBL surgical navigation prototype to function as the sole navigation system during spinal surgical procedures. The study will focus on testing the robustness of the system to appropriately function on a variety of spinal surgeries.

ELIGIBILITY:
Inclusion Criteria:

* Greater than 18 years of age, able to provide consent, or has substitute decision maker available to consent.
* Scheduled to undergo spinal instrumentation surgery involving pedicle or lateral mass screw insertion or brain tumor resection or biopsy.
* Scheduled for pre-operative CT/ MRI scan.
* No contra-indication for a post-operative CT/MRI scan.

Exclusion Criteria:

* Previous spinal decompression with significant laminectomy performed at the level intended for instrumentation
* Previous spinal decompression with laminoplasty performed at the level intended for instrumentation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-01-21 (Actual); Primary Completion 2019-01-21 (Estimated); Study Completion 2019-01-21 (Estimated)

PRIMARY OUTCOMES:
Pilot hole and screw trajectory accuracy as compared between post-operative CT and intraoperative images | Within 1 week of screw placement
  Comparison and quantification of accuracy of pilot holes including entry point and trajectory as taken from experimental navigation system as compared to absolute (or actual) entry point and trajectory of screws as determined by post-operative computed tomography scans.

CONTACTS AND LOCATIONS:
Overall Officials: Albert Yee, MD, MSc, Principal Investigator — Sunnybrook Health Sciences Centre; Victor XD Yang, MD, PhD, Principal Investigator — Sunnybrook Health Sciences Centre

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Merloz P, Tonetti J, Eld A, et al, Computer-assisted versus manual spine surgery: Clinical report, Springer Berlin, 1997.
- [Background] Rampersaud YR, Simon DA, Foley KT. Accuracy requirements for image-guided spinal pedicle screw placement. Spine (Phila Pa 1976). 2001 Feb 15;26(4):352-9. doi: 10.1097/00007632-200102150-00010. PMID 11224881
- [Background] Zdichaversusky M, Blauth M, Knop C, Graessner M, Herrmann H, Krettek C, Bastian L, Accuracy of Pedicle Screw Placement in Thoracic Spine Fractures, European Journal of Trauma, 30:234-240, 2004.
- [Background] Waters JD, Gonda DD, Reddy H, Kasper EM, Warnke PC, Chen CC. Diagnostic yield of stereotactic needle-biopsies of sub-cubic centimeter intracranial lesions. Surg Neurol Int. 2013 Apr 17;4(Suppl 3):S176-81. doi: 10.4103/2152-7806.110677. Print 2013. PMID 23682345
- [Background] Labadie RF, Davis BM, Fitzpatrick JM. Image-guided surgery: what is the accuracy? Curr Opin Otolaryngol Head Neck Surg. 2005 Feb;13(1):27-31. doi: 10.1097/00020840-200502000-00008. PMID 15654212
- [Background] Snyderman C, Zimmer LA, Kassam A. Sources of registration error with image guidance systems during endoscopic anterior cranial base surgery. Otolaryngol Head Neck Surg. 2004 Sep;131(3):145-9. doi: 10.1016/j.otohns.2004.03.002. PMID 15365528
- [Background] Pillai P, Sammet S, Ammirati M. Application accuracy of computed tomography-based, image-guided navigation of temporal bone. Neurosurgery. 2008 Oct;63(4 Suppl 2):326-32; discussion 332-3. doi: 10.1227/01.NEU.0000316429.19314.67. PMID 18981839
- [Background] Mathew JE, Mok K, Goulet B. Pedicle violation and Navigational errors in pedicle screw insertion using the intraoperative O-arm: A preliminary report. Int J Spine Surg. 2013 Dec 1;7:e88-94. doi: 10.1016/j.ijsp.2013.06.002. eCollection 2013. PMID 25694911
- [Background] Rajasekaran S, Vidyadhara S, Ramesh P, Shetty AP. Randomized clinical study to compare the accuracy of navigated and non-navigated thoracic pedicle screws in deformity correction surgeries. Spine (Phila Pa 1976). 2007 Jan 15;32(2):E56-64. doi: 10.1097/01.brs.0000252094.64857.ab. PMID 17224800